CLINICAL TRIAL: NCT00874744
Title: Phase 2 Study of Comparison of Single Intravitreal Injection of Triamcinolone or Bevacizumab for the Treatment of Diabetic Macular Edema.
Brief Title: Comparison of Single Intravitreal Injection of Triamcinolone or Bevacizumab for the Treatment of Diabetic Macular Edema
Acronym: Tribeva-DME
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade Federal de Goias (Other)
Responsible Party: David Leonardo Cruvinel Isaac, MD, Federal University of Goiás
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cerof-001
Record Dates: First submitted 2009-03-31; First posted 2009-04-02 (Estimated); Last update posted 2009-04-02 (Estimated); Status verified 2009-03

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic macular edema; intravitreal injection; Pharmacological treatment
MeSH Terms: interventions — Bevacizumab; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- bevacizumab (Experimental)
  Interventions: Drug: Bevacizumab
- Triamcinolone (Experimental)
  Interventions: Drug: Triamcinolone acetonide

INTERVENTIONS:
Drug: Bevacizumab — 1.25mg bevacizumab (0.05ml)
  Other Names: 1.Bevacizumab; 2.Avastin
  Arms: bevacizumab
Drug: Triamcinolone acetonide — 4.0 mg Triamcinolone acetonide injection
  Other Names: 1. Theracort; 2. Kenalog
  Arms: Triamcinolone

SUMMARY:
The purpose of this study is to compare a single intravitreal injection of 4.0 mg of triamcinolone acetonide and 1.25 mg of bevacizumab for the treatment of diabetic macular edema.

DETAILED DESCRIPTION:
Comparison a single intravitreal injection of 4.0 mg of triamcinolone acetonide and 1.25 mg of bevacizumab regarding the ability of central macular thickness reduction. Secondary objectives are analysis of Visual Outcomes and variations on Intraocular Pressure. The patients data were statistically analyzed if there was a 24 week follow up completed.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic macular edema with central foveal measurement over 300 micrometers

Exclusion Criteria:

* Glaucoma
* Vitreoretinal surgery
* Cataract Surgery less than 3 months prior inclusion
* Unilateral cataract surgery
* Uncontrolled Glycosylated Hemoglobin
* Previous Intraocular Injection
* Systemic Corticosteroids less than 1 month prior inclusion
* Macular ischemia at Fluorescein Angiography
* Cataract precluding fundus examination
* Active Proliferative Diabetic Retinopathy

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-03; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Comparison between the efficacy of a single intravitreal injection of 4.0mg of triamcinolone acetonide or 1.25mg of bevacizumab in the treatment of diabetic macular edema | 6 months

SECONDARY OUTCOMES:
To compare Visual Acuity between the same drug in Initial visit, 4, 12 ans 24 weeks and Visual Acuity between two group of eyes treated with different drugs. | 6 months
To compare Intraocular Pressure between the same drug in Initial visit, 4, 12 ans 24 weeks and Intraocular Pressure between two group of eyes treated with different drugs. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David LC Isaac, MD, PhD, Principal Investigator — Universidade Federal de Goias